CLINICAL TRIAL: NCT07074301
Title: Effectiveness of Education and Mobile Application for Percutaneous Endoscopic Gastrostomy Care
Brief Title: Training Program for PEG Caregivers: A Structured Intervention Study
Acronym: PEG-EDU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Sevilay Senol Celik, Professor of Nursing, Koç University School of Nursing, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024.389.IRB2.171
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Percutaneous Endoscopic Gastrostomy (PEG); Training; Caregiver Burden; Nutritional Support; Training Effectiveness
Keywords: Percutaneous endoscopic gastrostomy; Caregiver Burden; Structured Training; Home Enteral Nutrition
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel, randomized controlled trial involving caregivers of patients with PEG in Koç University Hospital. Participants will be randomly assigned to intervention (structured education and mobile application based on Bandura's Social Learning Theory) or control (routine care). Block randomization will be used, considering caregiver age and education level. Allocation concealment will be ensured via computer software. Data will be collected using standardized tools and analyzed independently to reduce bias.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor will be blinded to group assignments. Participants, care providers, and investigators will be aware of the intervention allocation due to the nature of the education and mobile application. Data analysis will be performed by an independent statistician to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver Training Program (Experimental): Caregivers receive a structured education program and mobile application support based on Bandura's Social Learning Theory.
  Interventions: Behavioral: Caregiver Training Program
- Routine Care (No Intervention): Caregivers receive the institution's standard information and support practices.

INTERVENTIONS:
Behavioral: Caregiver Training Program — The intervention consists of a two-month structured education program including two face-to-face sessions and a mobile application. The training content covers PEG care, stoma and tube management, enteral nutrition, drug administration via tube, and troubleshooting complications.
  Arms: Caregiver Training Program

SUMMARY:
This study aims to develop and evaluate a structured education program and a mobile application to support caregivers of patients receiving enteral nutrition via percutaneous endoscopic gastrostomy (PEG). The intervention focuses on improving caregivers' knowledge, care practices, and perceived burden. The study will be conducted in three phases: a needs assessment, development of the education and digital support modules, and implementation of the intervention. Quantitative and qualitative data will be collected to evaluate the impact of the intervention. The results are expected to contribute to the improvement of home PEG care quality and the empowerment of caregivers.

DETAILED DESCRIPTION:
This study is designed to improve the caregiving practices of individuals who are responsible for patients receiving long-term enteral nutrition via percutaneous endoscopic gastrostomy (PEG). The study is structured in three phases: (1) identification of caregivers' needs through descriptive and qualitative assessments, (2) development of a theory-based structured education program and a mobile application, and (3) implementation and evaluation of the intervention using a mixed-methods design.

In the first phase, caregivers' knowledge gaps, challenges, and educational needs will be identified through a needs assessment that includes questionnaires and semi-structured interviews. In the second phase, based on the findings of the initial assessment and supported by current clinical guidelines and national health policies, a structured education program and a digital support tool (mobile app) will be developed. The educational content will cover PEG fundamentals, stoma care, tube cleaning, enteral feeding, medication administration via PEG, complication management, and psychosocial support. Educational materials will include videos, animations, texts, and interactive quizzes, and the mobile app will allow asynchronous learning and monitoring.

In the third phase, the education program will be delivered through in-person theoretical and practical sessions, followed by the use of the mobile application. Outcome measures will include caregivers' knowledge level, caregiving burden, self-reported practices, and satisfaction with the intervention. Quantitative data will be collected using validated measurement tools, and qualitative feedback will be gathered to provide a deeper understanding of the intervention's impact. This study is expected to support the standardization of home PEG care and enhance caregiver capacity through sustainable and scalable educational interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willingness to participate voluntarily in the study
* No communication barriers
* Ability to use a smartphone
* No diagnosed psychiatric disorder
* Providing care to a patient aged 18 or older who is scheduled to undergo PEG placement

Exclusion Criteria:

* Discharge from hospital or death of the patient during the study period
* Being under 18 years old
* Illiteracy of the caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Caregiver Knowledge Level | Baseline and monthly assessments during 2-month intervention
  The effect of the training program and mobile application on the change in the knowledge level of caregivers (Data collection form to be used: Percutaneous Endoscopic Gastrostomy Care Knowledge Level Assessment Form). The form includes 28 items addressing PEG care (e.g., stoma care, tube maintenance, feeding, medication). Each correct answer scores 1 point. The total score ranges from 0 (lowest) to 28 (highest). Higher scores indicate greater knowledge.

SECONDARY OUTCOMES:
PEG Problems | Baseline and monthly assessments during 2-month intervention
  The impact of the training program and mobile app on the frequency and severity of PEG-related problems (blockage, infection, leakage, etc.) (Data collection form to be used: PEG Problems Monitoring Form). The form includes 12 predefined problem types (e.g., infection, leakage, dislodgement, constipation), and allows for open-ended documentation of additional complications. Each problem is recorded by date, severity (mild/moderate/severe), management approach, and outcome. Problems will be tracked monthly over a 2-month period. Higher number of recorded complications indicates a worse outcome.
Caregiver Burden Perception: | Baseline and monthly assessments during 2-month intervention
  The impact of the training program and mobile app on caregivers' perception of caregiver burden (Scale to be used: Zarit Caregiver Burden Scale). The Caregiver Burden Scale, a 21-item scale measuring the frequency of burden-related experiences. Each item is rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Almost always). Additionally, general caregiver stress is measured on a visual analogue scale from 0 (no stress) to 10 (extreme stress). Higher scores indicate a greater caregiver burden.
Training and Mobile Application Satisfaction: | Baseline and monthly assessments during 2-month intervention
  The user-friendliness of the training program and mobile application, and the level of satisfaction (Forms to be used: Training Evaluation Form, Mobile Application Evaluation Form, and Willingness to Use Mobile Application Scale). Caregiver satisfaction was assessed with the Training Evaluation Form (9 Likert-type items, score range: 9-45). Mobile app usability and content were explored via the Mobile Application Evaluation Form, including open-ended qualitative items. Willingness to use the app was measured by the Mobile Application Use Willingness Scale (6 items, 7-point Likert scale, total score: 6-42). Higher scores reflect greater satisfaction or willingness. Data were collected two months post-intervention.
Effectiveness of the Cleaning Brush | Baseline and monthly assessments during 2-month intervention
  Whether the cleaning brush is effective in maintaining PEG tubes and users' satisfaction with this product (Form to be used: Cleaning Brush Usage Evaluation Form).

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that supports the findings of this study will be available upon reasonable request from researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting documents (Study Protocol, SAP) will be available beginning 6 months after publication of the final results and will remain accessible for 3 years. Access will be granted upon reasonable request to the principal investigator.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access de-identified individual participant data (IPD), the study protocol, and the statistical analysis plan. Requests should be submitted to the principal investigator via institutional email and will be evaluated on a case-by-case basis. Data access will be granted through a secure institutional repository.